CLINICAL TRIAL: NCT06692127
Title: DETECTion of the Prevalence of Silent Atherosclerosis Across Adult Life and Development of a Risk Calculator to Predict Its Presence. Phase One of the REACT (Cure of Atherosclerosis) Project
Brief Title: DETECTion of the Prevalence of Silent Atherosclerosis Across Adult Life
Acronym: DETECT
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Novo Nordic Foundation (Other); Centro Nacional de Investigaciones Cardiovasculares Carlos III (Unknown); Gødstrup Hospital (Other); Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Henning Bundgaard, Professor of Cardiology, consultant, MD, DMSc, Rigshospitalet, Denmark
Other Study IDs: H-24047468
Record Dates: First submitted 2024-11-12; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Atheroslerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — Whole blood, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Atherosclerosis is preventable, yet it continues to significantly contribute to global morbidity and mortality. Atherosclerosis may occur early in life and may present in all vascular territories. The DETECT study's main aim is to determine the prevalence of asymptomatic atherosclerosis (silent) in an adult population of a wide age range of European ancestry through vascular ultrasound (VUS) of peripheral arteries (carotid and femoral territories), as well as establishing the relationship between atherosclerosis in peripheral arteries, coronary arteries, and other vascular territories assessed by computed tomography angiography (CTA).

The DETECT study also aims to identify risk factors for development of subclinical atherosclerosis that can hopefully improve the detection of the risk for development of atherosclerotic cardiovascular disease (ASCVD) with far higher precision than currently. In future research, the findings in this descriptive study may eventually be used as part of an age-adapted imaging-based screening for subclinical atherosclerosis.

The investigators hypothesize that a precision medicine-based approach to identify candidates likely to benefit from primary prevention against atherosclerosis, may improve medical decision making, by combining traditional risk factors, including lifestyle and psychological factors, phenotypic findings and findings on vascular imaging, and patterns of circulating biomarkers to identify risk of atherosclerosis especially in young individuals and at earlier disease stages (the ultimate population target of REACT project, phase II), maximizing the potential for prevention long before overt disease occurs. An essential aspect of this approach is to pinpoint the specific risk factors in each individual that primarily drive atherosclerosis throughout their life and could serve as therapeutic targets.

Thus, the overall purpose of this study is to establish the necessary knowledge, including extensive characterisation of atherosclerosis across life and thus add to the rational foundation for future development of a far more efficient and precise prophylaxis against ASCVD as compared with the presently applied methods.

ELIGIBILITY:
Inclusion Criteria:

* The study will include adults ≥18 to ≤70 years of age (1:1 sex ratio in each 10 years age strata).
* Have not been diagnosed with ASCVD prior to inclusion into the study (participants with other cardiovascular diseases or predisposing factors are not excluded).
* The participants will be recruited from sites in Denmark (n ~ 8,000) (and Spain (n ~ 8,000)).
* Participants need to be capable and be able to read and understand Danish, English, Spanish or Arabic.

Exclusion Criteria:

* The participants will be excluded from the CTA with contrast if they have severe renal disease (eGFR <30 ml), contrast allergies, pregnancy or other conditions excluding the performance of a CT-scan.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: spansk eog danske baggrundsbefolkning
Sampling Method: Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence of atherosclerosis | Immediately after the examination.
  Prevalence of atherosclerosis using imaging.

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (4):
  - Rigshospitalet, Copenhagen
  - Righospitalet - Glostrup Hospital, Glostrup Municipality
  - Herlev Hospital, Herlev
  - Regionshospitalet Gødstrup, Herning
- Centro Nacional de Investigaciones Cardiovasculares Carlos III (CNIC), Madrid, Spain

IPD SHARING:
Plan to Share IPD: No